CLINICAL TRIAL: NCT07199244
Title: The Immediate and Long-term Effects of Oral Administration of SalmoFer®, a Novel Marine-based Heme Iron Supplement, in Adult Females
Brief Title: The Immediate and Long-term Effects of a Novel Marine-based Iron Supplement in Adult Females
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Principal Investigator, Jessie Hawkins, Principal Investigator, Nutraceuticals Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-04-2500
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-01

CONDITIONS: Anemia; Iron Deficiency (Without Anemia); Iron Absorption
MeSH Terms: conditions — Anemia; Iron Deficiencies

STUDY DESIGN:
Masking Description: Participants are blinded to the dose and manufacturer of the supplement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplement Arm (Experimental): Individuals will consume the supplement for 56 days
  Interventions: Dietary Supplement: marine-based heme iron

INTERVENTIONS:
Dietary Supplement: marine-based heme iron — Participants will consume 9mg of SalmoFer on day 1, followed by 6mg each day for 56 days.

SUMMARY:
The goal of this study is to identify how well a fish-based iron supplement is absorbed and to learn how many, if any, digestive related side effects are caused by ingesting the supplement.

DETAILED DESCRIPTION:
This is a single population observational-style trial with a 24-hour pharmacokinetic evaluation. A minimum of 44 healthy adult female consented participants will be screened and classified as low-iron levels or anemic. Both classifications receive active iron supplements as a single group. Participants will provide data on the outcome measures of safety, vital signs, iron levels from whole blood collection, and subjective experience. Blood collection will take place at baseline, 30 minutes, 1 hour, 3 hours, 6 hours, 12 hours, and 24 hours after ingestion. All data will be taken at baseline and again at day 56, after daily intake of the supplement.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness and demonstrated ability to comply with all study procedures, as well as availability for the duration of the study
* Lives within 100 miles of a NRI study site
* Biological sex of woman; gender identification of female
* Aged 21 to 42, inclusive
* In luteal phase of menstrual cycle
* Either low levels of iron or mild-moderate iron-deficiency (defined as screening hemoglobin of 12.0-14.0 g/dL or 8.0-11.9 g/dL, respectively)
* Good general health as evidenced by medical history and screening metabolic panel and complete blood count (GMP & CBC)
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional month after the end of the study
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* A positive medical history of heart disease/cardiovascular disease, high blood pressure (140/90 or greater mmHg), kidney disease, hepatic impairment or disease, Type I or Type II diabetes, Irritable bowel disease/Irritable bowel syndrome (IBD/IBS), ulcerative colitis (UC), Crohn's disease or any other medical condition or diagnosis that the PI would deem exclusionary
* A positive surgical medical history for any procedure that may impact iron status (i.e., gastric bypass, gastric pull-up (Roux-en-Y), short bowel syndrome, etc
* A positive medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorder (i.e., HIV/AIDS), a history of cancer (except localized skin cancer without metastases or in situ cervical cancer within five years before the screening visit.
* A positive medical history of any gastrointestinal disease or illness
* A positive history of any other gastrointestinal surgery that is known to alter or impact the digestion absorption of nutrients and or fluids
* History of hospitalization or in-patient or out-patient treatment for alcohol dependence or drug addiction within the past two years
* History of hospitalization or in-patient treatment for depression or any related condition within the past five years
* Severe iron deficiency (defined as screening hemoglobin <8.0)
* Pregnancy, trying to conceive, or breastfeeding
* Currently smokes or vapes (i.e., tobacco, flavored items, marijuana, etc.) or has in the past year
* Known allergic reactions to any components of the intervention
* Positive COVID-19 test within 30 days of the study period
* Obese, defined as BMI >35
* Recent dramatic weight changes (10% change in body weight in the last 6 months)
* Existing usage of an iron supplement in any form
* Introducing a new investigational drug or other intervention within 60 days before the start of the study

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological sex of woman, gender of female
Enrollment: 61 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
total iron | baseline, 30min, 60 min, 3 hour, 6 hour, 12 hour, 24 hour, 56 days
  total iron measured through blood draws
Ferritin | baseline, 30min, 60 min, 3 hour, 6 hour, 12 hour, 24 hour, 56 days
  total ferritin assessed through blood draws
Transferrin | baseline, 30min, 60 min, 3 hour, 6 hour, 12 hour, 24 hour, 56 days
  transferrin measured through blood draws
hemoglobin | baseline, 30min, 60 min, 3 hour, 6 hour, 12 hour, 24 hour, 56 days
  hemoglogbin
hematocrit | baseline, 30min, 60 min, 3 hour, 6 hour, 12 hour, 24 hour, 56 days
  hematocrit measured through blood draws

SECONDARY OUTCOMES:
gastrointestinal discomfort | baseline, 30min, 3 hour, 6 hour, 24 hour, 56 days
  GI Discomfort is measured through a self-report scale which produces scores ranging from 1-5, with higher scores indicating higher levels of discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Nutraceuticals Research Institute, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
IPD may not be shared without a valid IRB authorization and consent of all study participants.